CLINICAL TRIAL: NCT03237013
Title: Strategies to Promote Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Aaron Blashill, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2253101
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Skin Cancer; Skin Cancer Melanoma; Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: Sunbathing; Indoor Tanning; Facial Morphing; Skin Cancer Risk
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Squamous Cell; Carcinoma, Basal Cell | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: At initial visit, participants were screened for study eligibility, consented, and randomized to a study condition. Participants first completed baseline assessment. Following, all participants completed intervention as determined by randomized assignment (i.e., control, facial morphing or mindfulness). At the initial visit, all subjects were assigned a subject ID number. Each subject ID was pre-assigned to a study condition, determined by an online randomization program, prior to recruitment. Each eligible participant had a 1/3 chance to be assigned to each of the three study conditions. Immediately after intervention, participants completed acute assessment, also consisting of self-report questionnaires. At the end of the initial visit, participants provided researchers a valid email address to be sent a subsequent follow-up survey. Approximately one month from the intervention date, participants received and completed the online follow-up survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Treatment as Usual only) (No Intervention): Following baseline assessment, all participants were given health literature on tanning behavior from the U.S. Centers for Disease Control and Prevention (CDC). These materials included informational pamphlets addressing common myths regarding tanning behaviors, including "Tanned skin is not healthy skin", and "A base tan is not a safe tan. These misconceptions were accompanied by "burning truth", scientific data debunking these myths. Additionally, all participants received a packet on sun protective practices for oneself and family, which include skin cancer statistics and information on UV rays.
- Treatment as Usual + Facial Morphing (Experimental): In addition to the health literature, participants completed the Facial Morphing Intervention. Participants had a digital photograph taken and uploaded to the APRIL® software, accompanied by information about their current age and self-identified race. Participants were presented with two, side-by-side identical 2D images of their face. Participants first viewed an image of their face from their current age, in two-year intervals, to age 72, the maximum age, with the "UV exposure" setting turned on. This process was repeated. Next, participants viewed the projected aging process, toggling the "UV exposure" setting (on and off), every ten year interval. The process was repeated using 3D images to view projected changes to their facial profiles.
  Interventions: Behavioral: Facial Morphing Intervention
- Treatment as Usual + Mindfulness (Placebo Comparator): In addition to the health literature, participants completed the Mindfulness Intervention. Participants listened to a 10-minute self-guided mindfulness audio exercise. The audio file is a scripted reading of an established, brief mindfulness exercise (Erisman & Roemer, 2010). During this guided session, participants learned what mindfulness was, when it can be used, and benefits from practice. Listeners were led through steps, focusing on the physical sensations, breathing, and thoughts. After the exercise, participants were provided a handout highlighting key points about mindfulness and how to incorporate informal mindfulness practice into their daily life.
  Interventions: Behavioral: Mindfulness Intervention

INTERVENTIONS:
Behavioral: Facial Morphing Intervention — Participants assigned to this condition were exposed to facial morphing technology that displays the progression of facial-ageing up to 72years, both with and without damage from UV exposure.
  Other Names: Facial Morphing
  Arms: Treatment as Usual + Facial Morphing
Behavioral: Mindfulness Intervention — Participants assigned to this condition engaged in a self-guided mindfulness intervention audio tape. This intervention instructed participants to pay attention to the present moment, with a non-judgemental stance. For example, participants were instructed to notice their breath, thoughts, feelings, physical sensations, and to internally describe them, without passing judgement
  Other Names: Mindfulness
  Arms: Treatment as Usual + Mindfulness

SUMMARY:
The purpose of the intended proposed research is to investigate and determine best strategies for preventing skin cancer for emerging adults. To answer this question, the investigators intended to pilot a randomized control trial with three arms: 1) Facial Morphing, 2) Mindfulness, and 3) Treatment as usual. The population from which the sample was drawn from was undergraduate psychology students from a large public university in Southern California, who report recent indoor/outdoor tanning, and intentions for future tanning.

DETAILED DESCRIPTION:
Indoor and outdoor tanning are two of the most common risk factors for developing skin cancer. Predictors of indoor and outdoor tanning including negative body image and negative affect. Thus, to subsequently prevent skin cancer, interventions should focus on appearance concerns and negative affect. To date, limited brief efficacious skin cancer preventions exist. One potential program (APRIL AGE) a facial morphing software program, has recently been evaluated as a potential prevention program of skin cancer. However, limited data exists on the long term benefits of this program. Additionally, brief mindfulness programs have been found to be efficacious in preventing other health risk behaviors (e.g., smoking, negative affect, eating behaviors). To the investigators' knowledge, these brief mindfulness interventions have yet to be applied in skin cancer prevention. Thus, the investigators sought to compare the relative efficacy of the facial morphing intervention and the mindfulness intervention vs. control condition (treatment as usual). It was hypothesized that both facial morphing and mindfulness would lead to reductions in tanning behavior compared to the TAU condition. The investigators also tested contrasts between the facial morphing and mindfulness conditions, however, no directional hypotheses could be generated, due to the dearth of prior data on these interventions in skin cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged 18 years old or older
* 2) enrolled as a student at the University
* 3) engaged in either indoor or outdoor tanning in the last 30 days
* 4) intended to tan (indoor or outdoor) in the last 30 days
* 5) English speaking

Exclusion Criteria:

* Failure to meet any of the above mentioned inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Blashill, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan at this time.

REFERENCES:
- [Background] Ashrafioun L, Bonar EE. Tanning addiction and psychopathology: Further evaluation of anxiety disorders and substance abuse. J Am Acad Dermatol. 2014 Mar;70(3):473-80. doi: 10.1016/j.jaad.2013.10.057. Epub 2013 Dec 25. PMID 24373775
- [Background] Ramos Diaz NS, Jimenez Jimenez O, Lopes PN. The role of mindfulness in coping with recollections of acute stressors: a laboratory study. Psicothema. 2014;26(4):505-10. doi: 10.7334/psicothema2014.71. PMID 25340898
- [Background] Erisman SM, Roemer L. A preliminary investigation of the effects of experimentally induced mindfulness on emotional responding to film clips. Emotion. 2010 Feb;10(1):72-82. doi: 10.1037/a0017162. PMID 20141304
- [Background] Hillhouse J, Stapleton J, Turrisi R. Association of frequent indoor UV tanning with seasonal affective disorder. Arch Dermatol. 2005 Nov;141(11):1465. doi: 10.1001/archderm.141.11.1465. No abstract available. PMID 16301398
- [Background] Marchiori D, Papies EK. A brief mindfulness intervention reduces unhealthy eating when hungry, but not the portion size effect. Appetite. 2014 Apr;75:40-5. doi: 10.1016/j.appet.2013.12.009. Epub 2013 Dec 20. PMID 24361312
- [Background] Rogojanski J, Vettese LC, Antony MM. Coping with cigarette cravings: Comparison of suppression versus mindfulness-based strategies. Mindfulness, 2(1): 14-26, 2011.
- [Background] Williams AL, Grogan S, Buckley E, Clark-Carter D. Men's experiences of an appearance-focussed facial-ageing sun protection intervention: a qualitative study. Body Image. 2013 Mar;10(2):263-6. doi: 10.1016/j.bodyim.2013.01.003. Epub 2013 Feb 9. PMID 23402802
- [Derived] Blashill AJ, Rooney BM, Luberto CM, Gonzales M 4th, Grogan S. A brief facial morphing intervention to reduce skin cancer risk behaviors: Results from a randomized controlled trial. Body Image. 2018 Jun;25:177-185. doi: 10.1016/j.bodyim.2018.04.002. PMID 29698824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted between February and December 2016. Participants were recruited from an undergraduate research participation website at a large, public American university. A general description of the study's purpose, which specified study inclusion criteria and one's time commitment was provided for potential participants
Groups:
- Treatment as Usual + Mindfulness: In addition to the health literature, participants completed the Mindfulness Intervention. Participants listened to a 10-minute self-guided mindfulness audio exercise. The audio file is a scripted reading of an established brief mindfulness exercise (Erisman & Roemer, 2010). During this guided session, participants learned what mindfulness was, when it can be used, and benefits from practice. Listeners were led through steps, focusing on the physical sensations, breathing, and thoughts. After the exercise, participants were provided a handout highlighting key points about mindfulness and how to incorporate informal mindfulness practice into their daily life.
  Mindfulness Intervention: Participants assigned to this condition engaged in a self-guided mindfulness intervention audio tape. This intervention instructed participants to pay attention to the present moment, with a non-judgemental stance. For example, participants were instructed to notice their breath, thoughts, feelings, ph
Period: Baseline to Immediate Post-treatment
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Started | 73 | 73 | 73
Completed | 73 | 73 | 73
Not Completed | 0 | 0 | 0
Period: Immediate Post-treatment to 1-mo F/u
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Started | 73 | 73 | 73
Completed (The number of participants who responded to the follow-up survey 1 month after intervention) | 30 | 43 | 36
Not Completed | 43 | 30 | 37
Not completed — Lost to Follow-up | 43 | 30 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness | Total
Number analyzed (Participants) | 73 | 73 | 73 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.60 (1.75) | 19.65 (2.77) | 19.90 (2.85) | 19.72 (2.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 64 | 57 | 178
  Male | 16 | 9 | 16 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 19 | 54
  Not Hispanic or Latino | 57 | 54 | 54 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 9 | 11 | 14 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 49 | 43 | 49 | 141
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 18 | 9 | 39
Region of Enrollment [Number; unit: participants]
  United States | 73 | 73 | 73 | 219
Skin Type [Count of Participants; unit: Participants] — Participants were asked to self-report their skin type among six options representing a range of light to dark skin tones indicating greater burning and tanning characteristics using the Fitzpatrick Skin Type Scale (Fitzpatrick, 1988). Participants were provided with six skin types (i.e., Skin Type I: Very Fair--always burns cannot tan; Skin Type 2: Fair--usually burns sometimes tans; Skin Type 3: Medium--sometimes burns usually tans; Skin Type 4: Olive--rarely burns always tans; Skin Type 5: Brown--never burns always tans; and Skin Type 6: Black--never burns always tans) to self-select from.
  Participants
    Skin Type I | 1 | 0 | 0 | 1
    Skin Type 2 | 10 | 9 | 6 | 25
    Skin Type 3 | 36 | 36 | 40 | 112
    Skin Type 4 | 23 | 24 | 27 | 74
    Skin Type 5 | 2 | 4 | 0 | 6
    Skin Type 6 | 1 | 0 | 0 | 1
Indoor Tanning Frequency [Mean (Standard Deviation); unit: Sessions in last month] — Participants reported the number of sessions of indoor tanning they experienced in the past month
  Sessions in last month | 1.30 (2.68) | 1.51 (2.83) | 1.28 (2.41) | 1.36 (2.62)
Outdoor Tanning Frequency [Mean (Standard Deviation); unit: Sessions in last month] — Participants were asked to self-report the number of sessions of outdoor tanning they engaged in within the last month
  Sessions in last month | 7.69 (5.35) | 7.25 (5.04) | 7.02 (4.84) | 7.32 (5.06)
Indoor Tanning Intentions [Mean (Standard Deviation); unit: Sessions in next month] — Participants were asked to estimate the number of times they plan to indoor tan in the next month
  Sessions in next month | 4.36 (2.17) | 4.13 (2.17) | 4.27 (2.20) | 4.25 (2.17)
Outdoor Tanning Intentions [Mean (Standard Deviation); unit: Sessions in next month] — Participants were asked to estimate the number of times they plan to outdoor tan in the next month
  Sessions in next month | 5.96 (1.37) | 5.56 (1.59) | 5.90 (1.20) | 5.81 (1.39)
Appearance Attitudes to Tan [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Appearance Reasons to Tan latent subscale of the Physical Appearance Reasons for Tanning Scale (PARTS; Cafri et al., 2006, 2008). This scale consists of three manifest subscales: General Attractiveness, Acne, and Body Shape. These 19 items were scored along a five-point scale: 1 (definitely disagree) to 5 (definitely agree), with a possible total score range of 19-95 (higher scores indicating greater agreement). Total scores are averaged to reflect the average agreement with attitudes which may motivate one to tan (higher average scores indicating greater agreement).
  units on a scale | 3.41 (0.76) | 3.29 (0.91) | 3.46 (0.74) | 3.42 (0.81)
Appearance Attitudes Not to Tan [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Appearance Reasons Not to Tan latent subscale of the Physical Appearance Reasons for Tanning Scale (PARTS; Cafri et al., 2006, 2008). This scale consists of two manifest subscales: Skin Damage and Skin Aging. These 9 items were scored along a five-point scale 1 (definitely disagree) to 5 (definitely agree) with a possible total score range of 9-45 (higher scores indicating greater agreement). Total scores are averaged to reflect the average agreement with attitudes to not tan; (higher average scores indicating greater agreement).
  units on a scale | 3.41 (0.76) | 3.31 (0.78) | 3.36 (0.77) | 3.36 (0.77)
State Body Satisfaction [Mean (Standard Deviation); unit: units on a scale] — State level body satisfaction was measured using the Body Image States Scale (BISS; Cash, Fleming, Alindogan, Steadman, & Whitehead, 2002). This six-item self-report instrument utilizes a nine-point scale (1 [extremely dissatisfied] to 9 [extremely satisfied]); possible total scores range 6-54; higher scores indicate greater satisfaction. This measure is scored by averaging all scores to these six items, with higher average scores indicating greater body satisfaction.
  units on a scale | 5.70 (1.35) | 5.48 (1.37) | 5.32 (1.37) | 5.50 (1.30)
Trait Body Satisfaction [Mean (Standard Deviation); unit: units on a scale] — Trait level body satisfaction was measured using the Multidimensional Body-Self Relations Questionnaire-Appearance Evaluation subscale (MSBRQ-AE; Brown, Cash, & Mikulka, 1990; Cash, 2000). This seven-item self-report subscale utilizes a five-point scale (1 [definitely disagree] to 5 [definitely agree]) with possible score range of 7-35. This measure was scored by averaging all scores to these seven items, with higher scores indicating greater body satisfaction.
  units on a scale | 3.52 (0.78) | 3.42 (0.68) | 3.39 (0.74) | 3.44 (0.73)
Appearance Orientation [Mean (Standard Deviation); unit: units on a scale] — Trait level appearance orientation satisfaction was measured using the Appearance Schemas Inventory-Revised Short Form (ASI-R; Cash, Melnyk, & Hrabosky, 2004). This twenty-item self-report instrument assesses cognitive and behavioral investment in one's physical appearance. This measure utilizes a five-point scale (1 [definitely disagree] to 5 [definitely agree]), with total scores ranging from 20-100; higher scores indicate greater appearance investment. This measure is scored by averaging all scores to these twenty items (higher scores indicating greater appearance investment).
  units on a scale | 3.66 (0.50) | 3.54 (0.58) | 3.64 (0.56) | 3.61 (0.55)
State Positive Affect [Mean (Standard Deviation); unit: units on a scale] — State positive affect was measured using the positive affect subscale of the Positive and Negative Affect Scale-Short Form (PANAS-SF; Thompson, 2007). This self-report subscale consists of five items of the full ten-item measure. This subscale utilizes a five-point Likert-type scale ranging from 1 (never) to 5 (always). This measure is scored by summing all scores to these five items (range 5-25), with higher scores indicating greater state positive affect. For the purposes of this project, participants' item scores to these five items were averaged.
  units on a scale | 3.59 (0.63) | 3.45 (0.76) | 3.33 (0.79) | 3.46 (0.74)
State Negative Affect [Mean (Standard Deviation); unit: units on a scale] — State negative affect was measured using the negative affect subscale of the Positive and Negative Affect Scale-Short Form (PANAS-SF; Thompson, 2007). This self-report subscale consists of five items of the full ten-item measure. This subscale utilizes a five-point Likert-type scale ranging from 1 (never) to 5 (always). This measure is scored by summing all scores to these five items (range 5-25), with higher scores indicating greater state negative affect. For the purposes of this project, participants' item scores to these five items were averaged.
  units on a scale | 2.20 (0.70) | 2.07 (0.75) | 2.02 (0.72) | 2.09 (0.72)
Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Depression Anxiety Stress Scales Short Version (DASS-21) as a marker of trait level negative affect (Henry & Crawford, 2005). This 21-item self-report measure consists of three seven-item subscales: depression, anxiety, and stress. Items are measured along a 4-point scale (0 [not at all like me] to 3 [applied to me very much, or most of the time]); higher scores denote increased symptoms. Total sum scores for this instrument ranges from 0-63; scores for the depressive symptom subscale range from 0-21.
  units on a scale | 4.82 (4.95) | 6.32 (8.84) | 5.97 (7.59) | 5.70 (7.30)
Anxiety Symptoms [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Depression Anxiety Stress Scales Short Version (DASS-21) as a marker of trait level negative affect (Henry & Crawford, 2005). This 21-item self-report measure consists of three seven-item subscales: depression, anxiety, and stress. Items are measured along a 4-point scale (0 [not at all like me] to 3 [applied to me very much, or most of the time]); higher scores denote increased symptoms. Total sum scores for this instrument ranges from 0-63; scores for the anxiety symptom subscale range from 0-21.
  units on a scale | 6.63 (5.82) | 7.86 (7.83) | 6.38 (5.86) | 6.95 (6.57)
Stress [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Depression Anxiety Stress Scales Short Version (DASS-21) as a marker of trait level negative affect (Henry & Crawford, 2005). This 21-item self-report measure consists of three seven-item subscales: depression, anxiety, and stress. Items are measured along a 4-point scale (0 [not at all like me] to 3 [applied to me very much, or most of the time]); higher scores denote increased symptoms. Total sum scores for this instrument ranges from 0-63; scores for the stress symptom subscale range from 0-21.
  units on a scale | 10.38 (7.82) | 11.39 (9.28) | 11.56 (8.82) | 11.11 (8.63)

OUTCOME MEASURES:

1. Primary Outcome: Number of Indoor Tanning Sessions in the Last 30 Days
Description: One free-response item measuring intentional indoor frequency in the last 30 days
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: Sessions in last month
Groups:
- Treatment as Usual + Mindfulness: In addition to the health literature, participants completed the Mindfulness Intervention. Participants listened to a 10-minute self-guided mindfulness audio exercise. The audio file is a scripted reading of an established, brief mindfulness exercise (Erisman & Roemer, 2010). During this guided session, participants learned what mindfulness was, when it can be used, and benefits from practice. Listeners were led through steps, focusing on the physical sensations, breathing, and thoughts. After the exercise, participants were provided a handout highlighting key points about mindfulness and how to incorporate informal mindfulness practice into their daily life.
  Mindfulness Intervention: Participants assigned to this condition engaged in a self-guided mindfulness intervention audio tape. This intervention instructed participants to pay attention to the present moment, with a non-judgemental stance.
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
Sessions in last month | 1.98 (3.21) | 1.35 (2.81) | 1.92 (2.86)

2. Primary Outcome: Number of Outdoor Tanning Sessions in the Last 30 Days
Description: One free-response item measuring intentional outdoor frequency in the last 30 days
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: Sessions in last month
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
Sessions in last month | 3.96 (4.07) | 2.69 (3.31) | 3.24 (3.60)

3. Primary Outcome: Indoor Tanning Intentions
Description: A free-response items measuring intentional indoor intentions in the next 30 days.
Time Frame: Post assessment & 1-month assessment
Measure: Mean (Standard Deviation); unit: sessions in next month
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
sessions in next month
  Post-Assessment | 3.10 (2.05) | 2.21 (1.59) | 2.74 (2.07)
  1-Month Assessment | 3.12 (1.90) | 2.60 (1.76) | 3.16 (1.82)

4. Primary Outcome: Outdoor Tanning Intentions
Description: A free-response items measuring intentional outdoor intentions in the next 30 days.
Time Frame: Post Assessment & 1-month assessment
Measure: Mean (Standard Deviation); unit: sessions in next month
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
sessions in next month
  Post-Assessment | 4.53 (1.74) | 3.41 (1.85) | 4.53 (1.62)
  1-Month Assessment | 3.48 (1.97) | 3.37 (1.83) | 3.89 (1.76)

5. Secondary Outcome: Appearance Attitudes to Tan
Description: Participants completed the Appearance Reasons to Tan latent subscale of the Physical Appearance Reasons for Tanning Scale (PARTS; Cafri et al., 2006, 2008). This scale consists of three manifest subscales: General Attractiveness, Acne, and Body Shape. These 19 items were scored along a five-point scale: 1 (definitely disagree) to 5 (definitely agree), with a possible total score range of 19-95 (higher scores indicating greater agreement). Total scores are averaged to reflect the average agreement with attitudes which may motivate one to tan (higher average scores indicating greater agreement).
Time Frame: Post assessment & 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale
  Post-assessment | 3.28 (0.90) | 2.90 (0.99) | 3.25 (0.76)
  1-Month Assessment | 3.22 (0.66) | 3.13 (0.80) | 3.13 (0.61)

6. Secondary Outcome: Appearance Reasons Not to Tan
Description: Participants completed the Appearance Reasons Not to Tan latent subscale of the Physical Appearance Reasons for Tanning Scale (PARTS; Cafri et al., 2006, 2008). This scale consists of two manifest subscales: Skin Damage and Skin Aging. These 9 items were scored along a five-point scale 1 (definitely disagree) to 5 (definitely agree) with a possible total score range of 9-45 (higher scores indicating greater agreement). Total scores are averaged to reflect the average agreement with attitudes to not tan; (higher average scores indicating greater agreement).
Time Frame: Post assessment and 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale
  Post-Assessment | 3.74 (0.79) | 3.83 (0.93) | 3.63 (0.83)
  1-Month Assessment | 3.40 (0.72) | 3.61 (0.82) | 3.59 (0.62)

7. Secondary Outcome: State Body Satisfaction
Description: State level body satisfaction was measured using the Body Image States Scale (BISS; Cash, Fleming, Alindogan, Steadman, & Whitehead, 2002). This six-item self-report instrument utilizes a nine-point scale (1 [extremely dissatisfied] to 9 [extremely satisfied]); possible total scores range 6-54; higher scores indicate greater satisfaction. This measure is scored by averaging all scores to these six items, with higher average scores indicating greater body satisfaction.
Time Frame: Post-assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 5.67 (1.28) | 5.36 (1.41) | 5.49 (1.34)

8. Secondary Outcome: Trait Body Satisfaction
Description: Trait level body satisfaction was measured using the Multidimensional Body-Self Relations Questionnaire-Appearance Evaluation subscale (MSBRQ-AE; Brown, Cash, & Mikulka, 1990; Cash, 2000). This seven-item self-report subscale utilizes a five-point scale (1 [definitely disagree] to 5 [definitely agree]) with possible score range of 7-35. This measure was scored by averaging all scores to these seven items, with higher scores indicating greater body satisfaction.
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 3.32 (0.68) | 3.33 (0.66) | 3.30 (0.70)

9. Secondary Outcome: Appearance Orientation
Description: Trait level appearance orientation satisfaction was measured using the Appearance Schemas Inventory-Revised Short Form (ASI-R; Cash, Melnyk, & Hrabosky, 2004). This twenty-item self-report instrument assesses cognitive and behavioral investment in one's physical appearance. This measure utilizes a five-point scale (1 [definitely disagree] to 5 [definitely agree]), with total scores ranging from 20-100; higher scores indicate greater appearance investment. This measure is scored by averaging all scores to these twenty items (higher scores indicating greater appearance investment).
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 3.50 (0.47) | 3.34 (0.49) | 3.42 (0.44)

10. Secondary Outcome: State Positive Affect
Description: State positive affect was measured using the positive affect subscale of the Positive and Negative Affect Scale-Short Form (PANAS-SF; Thompson, 2007). This self-report subscale consists of five items of the full ten-item measure. This subscale utilizes a five-point Likert-type scale ranging from 1 (never) to 5 (always). This measure is scored by summing all scores to these five items (range 5-25), with higher scores indicating greater state positive affect. For the purposes of this project, participants' item scores to these five items were averaged.
Time Frame: Post assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 3.45 (0.82) | 3.32 (0.92) | 3.31 (0.80)

11. Secondary Outcome: State Negative Affect
Description: State negative affect was measured using the negative affect subscale of the Positive and Negative Affect Scale-Short Form (PANAS-SF; Thompson, 2007). This self-report subscale consists of five items of the full ten-item measure. This subscale utilizes a five-point Likert-type scale ranging from 1 (never) to 5 (always). This measure is scored by summing all scores to these five items (range 5-25), with higher scores indicating greater state negative affect. For the purposes of this project, participants' item scores to these five items were averaged.
Time Frame: Post assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 1.95 (0.73) | 2.22 (0.80) | 1.72 (0.77)

12. Secondary Outcome: Depressive Symptoms
Description: Participants completed the Depression Anxiety Stress Scales Short Version (DASS-21) as a marker of trait level negative affect (Henry & Crawford, 2005). This 21-item self-report measure consists of three seven-item subscales: depression, anxiety, and stress. Items are measured along a 4-point scale (0 [not at all like me] to 3 [applied to me very much, or most of the time]); higher scores denote increased symptoms. Total sum scores for this instrument ranges from 0-63; scores for the depressive symptom subscale range from 0-21.
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 11.35 (7.91) | 9.16 (8.00) | 12.06 (8.56)

13. Secondary Outcome: Anxiety Symptoms
Description: Participants completed the Depression Anxiety Stress Scales Short Version (DASS-21) as a marker of trait level negative affect (Henry & Crawford, 2005). This 21-item self-report measure consists of three seven-item subscales: depression, anxiety, and stress. Items are measured along a 4-point scale (0 [not at all like me] to 3 [applied to me very much, or most of the time]); higher scores denote increased symptoms. Total sum scores for this instrument ranges from 0-63; scores for the anxiety symptom subscale range from 0-21.
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 13.22 (8.40) | 10.74 (8.63) | 12.82 (8.81)

14. Secondary Outcome: Stress
Description: Participants completed the Depression Anxiety Stress Scales Short Version (DASS-21) as a marker of trait level negative affect (Henry & Crawford, 2005). This 21-item self-report measure consists of three seven-item subscales: depression, anxiety, and stress. Items are measured along a 4-point scale (0 [not at all like me] to 3 [applied to me very much, or most of the time]); higher scores denote increased symptoms. Total sum scores for this instrument ranges from 0-63; scores for the stress symptom subscale range from 0-21.
Time Frame: 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
Number analyzed (Participants) | 30 | 43 | 36
units on a scale | 16.75 (9.29) | 14.02 (9.02) | 15.43 (8.96)

ADVERSE EVENTS:
Time Frame: 11 months
Description: Adverse events were monitored/assessed, however, no adverse events occurred/were reported to study personnel. No adverse events to report.
Arm/Group | Control (Treatment as Usual Only) | Treatment as Usual + Facial Morphing | Treatment as Usual + Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes